CLINICAL TRIAL: NCT05776836
Title: A Prospective and Multicentric Investigation Evaluating the Clinical Safety of FASY F and FASY P Hyaluronic Acid Gel for the Treatment of Pathological Facial Lipoatrophy
Brief Title: Evaluation of HA Dermal Fillers in the Treatment of Pathological Facial Lipoatrophy
Acronym: HAtrophy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Symatese (Industry)
Collaborators: EVAMED (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CLIN2203
Record Dates: First submitted 2023-02-24; First posted 2023-03-20 (Actual); Last update posted 2025-03-13 (Actual); Status verified 2025-03

CONDITIONS: Facial Lipoatrophy (FLA)
Keywords: Hyaluronic acid; Dermal fillers; Lipoatrophy
MeSH Terms: conditions — Lipodystrophy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- FASY (Experimental): Subjects will be consecutively included to receive FASY F in cheeks and nasolabial folds and FASY P in periorbital areas.
  Interventions: Device: Dermal filler

INTERVENTIONS:
Device: Dermal filler — Subjects will be consecutively included to receive FASY F in nasolabial folds and cheeks and FASY P in periorbital areas.

SUMMARY:
Facial lipoatrophy (FLA) refers to the loss of adipose tissue and is manifested by flattening or indentation of convex contours of the face. Most frequently, the subcutaneous layer is affected and most common locations of adipose tissue loss are the cheeks, temples, preauricular, orbital or perioral and oral areas. Most common etiology for FLA is related to HIV. In 1998, first FLA was described in Subjects under highly active antiretroviral therapy (HAART). Currently, no specific treatment for FLA is known. For HIV-associated FLA, the European AIDS Clinical Society (EACS) recommends in prevention, the avoidance of some ART (Active Antiretroviral therapy) such as stavudine and zidovudine. In corrective purpose, the switch of ART is advisable as well as surgical intervention involving dermal fillers.

Different filling treatment options are available to treat volume defect on FLA Subjects including PolyLactic Acid (PLLA) (i.e.; Sculptra®), Calcium hydroxyapatite ( CaHa - i.e.: Radiesse®), autologous fat graft and hyaluronic acid (HA). Several studies shown promising results for the use of HA in this indication with good reconstructive and aesthetic outcomes, excellent safety profile and comparable to the autologous fat transfer treatment. HA fillers are described as voluming agents for treatment of FLA associated with fat wasting disorders, lasting at least 6 months but the persistent volumetric effect depends on HA crosslinking level and concentration.

DETAILED DESCRIPTION:
The study is a pilot, prospective, multicenter, proof-of-concept clinical trial that aims to evaluate the safety and efficacy of FASY F and FASY P products for the treatment of FLA.

ELIGIBILITY:
Inclusion Criteria:

1. Sex: male or female.
2. Age: 18 years and older.
3. If female of child-bearing potential, must have a negative urine pregnancy test before the first injection and use a reliable form of contraception for more than 12 weeks prior to screening and throughout the investigation.

   Note: to be considered females of non-child-bearing potential, females must be surgically sterile or postmenopausal or under highly effective birth control methods as: combined hormonal contraception (containing estrogens and progestogen) associated with inhibition of ovulation (oral, intravaginal, transdermal); progestogen only hormonal contraception associated with inhibition of ovulation (oral, injectable, implantable); intrauterine device (IUD); intrauterine hormone-releasing system (IUS); bilateral tubal occlusion; vasectomized partner; sexual abstinence documented in medical history for at least 1 year.
4. In case of HIV:

   * HIV infection with a non-detectable viral charge (viral load <50 copies/mL) confirmed by a recent blood analysis.
   * Patient with platelet count greater than 50,000 cells/L by a recent blood analysis.
5. Patient with mild to moderate facial lipoatrophy based on "Ascher lipoatrophy Scale" scale (grade II to IV).
6. Patient, having given freely and expressly his/her informed consent.
7. Patient who is able to comply with the study requirements, as defined in the present clinical investigation protocole, at the Investigator's appreciation.
8. Patient being affiliated to a health social security system.

Exclusion Criteria:

1. Pregnant and breastfeeding women
2. Subject who is deprived of their freedom by administrative or legal decision.
3. Subject living in a social or sanitary establishment.
4. Major subject who is under guardianship or who is not able to express his consent.
5. Subject being in an exclusion period for a previous study or with a current or recent (<3 months) participation in another investigational study involving a drug or combined device with drug.
6. Subject who has scars, moles, sunburn, too many hairs, or other blemishes in the test area (face) which would interfere with the evaluation.
7. Subject suffering from a severe or progressive disease or any other pathology that may interfere with the evaluation of the study results: diabetes, autoimmune pathology, cardiac pathologies, hepatic deficiency, epilepsy, porphyria (other than HIV and related HIV disease).
8. Subject who has a known history of severe multiple allergies, angioedema or anaphylactic shock.
9. Subject with a known allergy or hypersensitivity to Hyaluronic Acid or local anesthesia (Lidocaine or anesthetics of the amide type or any of the excipients)
10. Subject with an acute inflammatory process or active skin disease, or related conditions, such as infection, psoriasis, rosacea, acne, blotches or other pathology near or on the injection sites with the potential to interfere with the study results or increase the risk of Adverse Events at the Investigator appreciation (other than HIV and related HIV disease).
11. Subject with a past history of severe streptococcal disease or an active streptococcus infection.
12. Subject predisposed to keloid or hypertrophic scarring.
13. Subject with a disorder that may impact wound healing such as connective tissue or immunosuppressive disorder (other than HIV and related HIV disease).
14. Subject with a history of precancerous lesions/skin malignancies on the injection sites.
15. Subject with history of hyper- or hypo-pigmentation on the face.
16. Subject with a known bleeding disorder or receiving medication that will likely increase the risk of bleeding during treatment, at the Investigator appreciation.
17. Subject having received high dose of Lidocaine (more than 200mg) and/or high dose of anesthetics structurally related to amide-type within the past week.
18. Subject having received chemotherapy agents, immunosuppressive medications or systemic corticosteroids within the past 3 months.
19. Patient having taken high-dose aspirin, anti-inflammatories, antiplatelet, thrombolytic during the week before the injection session.
20. Subject having received within the past 12 months any injections including nonpermanent fillers (e.g., Hyaluronic Acid, CaHA), mesotherapy or neurotoxin near or on the cheeks and/or cheekbones and/or infraorbital hollows or plan to undergo such treatment during the study.
21. Subject with prior permanent implant or treatment with non-HA or non-collagen filler near or on the cheeks and/or cheekbones and/or infraorbital hollows or plan to implement these products at any time during the study.
22. Subject having received within the past 6 months mesotherapy, resurfacing laser, photo modulation, intense pulsed light, radio frequency, photo-rejuvenation, dermabrasion, chemical peel, or other ablative or none ablative procedures near or on cheekbones and/or infraorbital hollows.
23. Subject with subcutaneous retaining structure on the face (meshing, threads, gold strand etc.).
24. Patient having received fat grafting within the past 12 months
25. Other condition preventing the subject to participate the study in the Investigator's opinion: subject deemed unreliable or incapable of understanding and complying with the study assessment or unrealistic expectations of treatment results.
26. Subject willing to perform any aesthetic treatment on the face other than treatment planned in the protocol during the study period.
27. Subject who have planned an intensive exposure to sunlight or UV-rays in the 2 weeks following injection.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2023-08-28 (Actual); Primary Completion 2023-12-13 (Actual); Study Completion 2024-11-26 (Actual)

PRIMARY OUTCOMES:
Proportion of subjects with at least one Injection Site Reaction within 30 days after the last injection. | 30 days visit after the last injection.
  Recording of the occurrence of local injection site reactions for each injection areas (cheeks, nasolabial folds, periorbital). Assessed by investigators.

SECONDARY OUTCOMES:
Injection Site Reactions present within the 14 days of the last injection. | During 14 days after the last injection.
  Recording in a daily diary of the presence and severity of local injection site reactions for each injection areas (cheeks, nasolabial folds, periorbital). Assessed by patients.
Global safety evaluation | Day 30, Month 3, Month 6, Month 9 and Month 12 after the last injection.
  Collection of Adverse Event assessed and recorded by investigators.
Visual analogic scale pain assessment. | Immediately after the injection (for initial injection only)
  Description: Assessment of pain using a 0-100mm Visual Analogue Scale for each injection area. (0 corresponds to no pain and 100 corresponds to the highest pain that can be felt).
Lipoatrophy severity modification | Baseline, Day 30, Month 3, Month 6, Month 9 and Month 12 after the last injection.
  Assessemnt of the level of facial lipoatrophy using Ascher Lipoatrophy Scale, a 5-point scale ranking from grade 1: Mild flattening or shadowing of one or more facial regions to grade 5: Severe indentation of one or more facial regions. The lower the score, the better the aesthetic result. Assessed by investigators.
Facial volume quantification | Baseline, Day 30, Month 3, Month 6, Month 9 and Month 12 after the last injection.
  Quantitative measure of cheeks, nasolabial fold and infraorbital hollows volumes (in milliliter) measured using Quantificare® program based on 3D LIFEVIZ mini® photographs.
Quality of life assessement | Day 30, Month 3, Month 6, Month 9 and Month 12 after the last injection.
  Assessment of patient's quality of life using the Facial Appearance Inventory scale, a 7-grade scale ranking from 1:very negative to 7: very positive. The higher the score, the better the quality of life. Assessed by patients.
Patient Global aesthetic improvement | Before touch-up, if any, then at Day 30, Month 3, Month 6, Month 9 and Month 12 after the last injection..
  Aesthetic improvement of the face will be assessed using the Global Aesthetic Improvement Scale, a 5-point scale ranking from 1: Very much improved to 5: worse. The lower the score, the better the aesthetic result. Assessed by subjects.
Investigator Global aesthetic improvement | Before touch-up, if any, then at Day 30, Month 3, Month 6, Month 9 and Month 12 after the last injection.
  Aesthetic improvement of the face will be assessed using the Global Aesthetic Improvement Scale, a 5-point scale a 5-point scale ranking from 1: Very much improved to 5: worse. The lower the score, the better the aesthetic result. Assessed by investigators.
Implant card readability. | Day 0
  Assessment of the reading and understanding of the FASY F or FASY P implant card by 15 subjects using a questionnaire on which the text present on the implant card must be identified and reported.

CONTACTS AND LOCATIONS:
Locations (3):
- France (3):
  - Palais de Flore, Lyon, Rhone
  - THINKIN, Paris, Île-de-France Region
  - Dermatology practice, Saint-Maur-des-Fossés, Île-de-France Region

IPD SHARING:
Plan to Share IPD: No